CLINICAL TRIAL: NCT06353256
Title: Alabama Womb 2 Heart Solution (AW2H): A Community Health Worker Intervention to Improve Short- and Long-term Outcomes in Black Patients With Adverse Pregnancy Outcomes
Brief Title: A Community Health Worker Intervention to Address Adverse Pregnancy Outcomes
Acronym: AW2H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Heart Association (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jesse Rattan, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300012607; 24POST1198805 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2024-03-28; First posted 2024-04-09 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Preeclampsia Postpartum; Adverse Pregnancy Outcomes
Keywords: community health workers; adverse pregnancy outcomes; preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Experimental): Usual postpartum care
  Interventions: Behavioral: usual postpartum care
- Usual care and community health worker intervention (Experimental): Usual postpartum care and community health worker visits and support
  Interventions: Behavioral: usual postpartum care + community health worker intervention

INTERVENTIONS:
Behavioral: usual postpartum care — Usual clinical and educational postpartum care
  Arms: Usual Care
Behavioral: usual postpartum care + community health worker intervention — participants will receive routine care and also community health worker support and visits.
  Arms: Usual care and community health worker intervention

SUMMARY:
United States maternal mortality and preterm birth rates are among the highest among high-income countries due in part to a combination of racial, regional and socioeconomic disparities in access to care and overall health. The research proposed focuses on adapting and expanding a perinatal community health worker intervention for Black postpartum patients with preeclampsia (PE) and other adverse pregnancy outcomes (APOs). Investigators will partner with a community-based organization that trains and deploys community health workers. Investigators will test an intervention for urban and rural Black postpartum patients with APOs to 1) enhance blood pressure control postpartum and 2) promote long-term cardiovascular disease prevention for this underserved population. This pilot study will determine if randomizing and implementing a community health worker intervention tailored to pregnant people experiencing preeclampsia is feasible and found to be acceptable by participants.

DETAILED DESCRIPTION:
The investigators will adapt a current perinatal community health worker intervention, lead by a leading community health worker organization, Connection Health, to the unique needs of Black postpartum patients with preeclampsia and other adverse pregnancy outcomes. The investigators will conduct a pilot trial to assess the feasibility and acceptability of the intervention. The hypothesis is that it is possible to randomize eligible patients to the feasibility trial, and the intervention will be acceptable to participants. The investigators will randomize Black postpartum patients with preeclampsia or other adverse pregnancy outcomes to either 1) usual care - cardiovascular disease-prevention education before discharge, or 2) intervention - cardiovascular disease prevention education before discharge plus an adapted Connection Health community health worker intervention. Following the completion of this project, the investigators intend to conduct a larger postpartum community health worker intervention trial in patients with preeclampsia or other adverse pregnancy outcomes powered to detect a difference in clinically meaningful outcomes, as informed by our existing community advisory board.

ELIGIBILITY:
Inclusion Criteria:

* Self Identifies as Black
* Between 16-56 years old
* Experiencing adverse pregnancy outcomes defined as hypertensive disorders of pregnancy, preterm birth, placental abruption, pregnancy loss (loss at greater or equal to 14 weeks gestation), gestational diabetes, delivering a small for gestational age infant
* Planning to deliver at UAB Hospital
* Speaks and writes in English

Exclusion Criteria:

* Declines Randomization
* Speaks or writes in languages other than English
* Currently incarcerated
* Previously enrolled in P3OPPY

Ages: 16 Years to 56 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Acceptability | 12 weeks
  Participant satisfaction with postpartum support received as part of the study (scaled from 1 to 10).

SECONDARY OUTCOMES:
Patient satisfaction with CHW intervention | 6-12 weeks postpartum
  Patient satisfaction with CHW intervention using Sekhon Questionnaire to Assess the Acceptability of Healthcare Interventions, 1-5 scale with 1 being the lowest acceptability to 5 being the highest acceptability.
Secondary Outcome Measure: Primary Care Visit Scheduled | 6-12 weeks postpartum
  Participant reports at least one visit is scheduled with a primary care provider
Secondary Outcome Measure: Mean Blood Pressure | 6-12 weeks postpartum
  Mean blood pressure at 6-12 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Jesse E Rattan, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - UAB Medicine, Birmingham, Alabama
  - The University of Alabama at Birmingham, Birmingham, Alabama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention.Maternal Mortality by State, 2018. US Department of Health and Human Services. National Center for Health Statistics.
- [Background] Parikh NI, Gonzalez JM, Anderson CAM, Judd SE, Rexrode KM, Hlatky MA, Gunderson EP, Stuart JJ, Vaidya D; American Heart Association Council on Epidemiology and Prevention; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular and Stroke Nursing; and the Stroke Council. Adverse Pregnancy Outcomes and Cardiovascular Disease Risk: Unique Opportunities for Cardiovascular Disease Prevention in Women: A Scientific Statement From the American Heart Association. Circulation. 2021 May 4;143(18):e902-e916. doi: 10.1161/CIR.0000000000000961. Epub 2021 Mar 29. PMID 33779213
- [Background] Leitao S, Manning E, Greene RA, Corcoran P; Maternal Morbidity Advisory Group*. Maternal morbidity and mortality: an iceberg phenomenon. BJOG. 2022 Feb;129(3):402-411. doi: 10.1111/1471-0528.16880. Epub 2021 Sep 23. PMID 34455672
- [Background] Minehart RD, Bryant AS, Jackson J, Daly JL. Racial/Ethnic Inequities in Pregnancy-Related Morbidity and Mortality. Obstet Gynecol Clin North Am. 2021 Mar;48(1):31-51. doi: 10.1016/j.ogc.2020.11.005. PMID 33573789
- [Background] Garovic VD, Dechend R, Easterling T, Karumanchi SA, McMurtry Baird S, Magee LA, Rana S, Vermunt JV, August P; American Heart Association Council on Hypertension; Council on the Kidney in Cardiovascular Disease, Kidney in Heart Disease Science Committee; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Lifestyle and Cardiometabolic Health; Council on Peripheral Vascular Disease; and Stroke Council. Hypertension in Pregnancy: Diagnosis, Blood Pressure Goals, and Pharmacotherapy: A Scientific Statement From the American Heart Association. Hypertension. 2022 Feb;79(2):e21-e41. doi: 10.1161/HYP.0000000000000208. Epub 2021 Dec 15. PMID 34905954